CLINICAL TRIAL: NCT03410043
Title: Randomized Phase II Trial of Osimertinib With or Without Local Consolidation Therapy (LCT) for Patients With EGFR-Mutant Metastatic NSCLC (NORTHSTAR)
Brief Title: Osimertinib, Surgery, and Radiation Therapy in Treating Patients With Stage IIIB or IV Non-small Cell Lung Cancer With EGFR Mutations, NORTHSTAR Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0228; NCI-2018-00937 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0228 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IIIB Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — osimertinib; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (LCT) (Experimental): Patients receive osimertinib PO QD for 6-12 weeks. Patients then undergo surgery and/or radiation therapy daily for 5 consecutive days every week for up to 8 weeks. Patients continue osimertinib during and after radiation therapy. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Osimertinib; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery
- Group II (no LCT) (Experimental): Patients receive osimertinib PO QD. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Given PO
  Other Names: AZD-9291; AZD9291; Mereletinib; Tagrisso
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Group I (LCT)
Procedure: Therapeutic Conventional Surgery — Undergo surgery
  Arms: Group I (LCT)

SUMMARY:
This phase II trial studies how well osimertinib, surgery, and radiation therapy work in treating patients with stage IIIB or IV non-small cell lung cancer with EGFR mutations. Osimertinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving osimertinib, surgery, and radiation therapy may work better at treating non-small cell lung cancer with EGFR mutations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether, in patients with tyrosine kinase inhibitor (TKI) naive or TKI resistant (acquired T790M) metastatic EGFR mutant non-small cell lung cancer (NSCLC) who do not progress after 6-12 weeks of induction osimertinib, local consolidative therapy (LCT; radiotherapy +/- surgical resection) followed by osimertinib prolongs progression-free survival (PFS) compared with osimertinib alone.

SECONDARY OBJECTIVES:

I. To determine whether osimertinib plus LCT improves time to progression of non-irradiated lesions (TTP-NIL) and time to appearance of new metastases (TANM) compared with osimertinib alone.

II. To determine whether osimertinib plus LCT improves the time to progression of target versus (vs.) non-target lesions compared with osimertinib alone.

III. To determine whether osimertinib plus LCT improves progression-free survival compared with osimertinib alone in TKI naive EGFR (L8585R/exon 19 deletion) mutant metastatic NSCLC.

IV. To determine whether osimertinib plus LCT improves progression-free survival compared with osimertinib alone in TKI resistant (acquired T790M) EGFR mutant NSCLC.

V. To determine whether osimertinib plus LCT improves progression-free survival compared with osimertinib alone in the subgroup of patients with oligometastatic NSCLC (up to 3 metastases).

VI. To assess the safety and tolerability of osimertinib with and without LCT. VII. To determine whether osimertinib plus LCT improves overall survival (OS) compared with osimertinib alone.

VIII. To determine if there is a difference in survival outcomes or toxicity by radiation treatment modality (protons vs. photons).

EXPLORATORY OBJECTIVES:

I. To explore the association of baseline genomic, proteomic and gene expression profiles (from tumor, germline deoxyribonucleic acid [DNA], and cell free [cf]DNA) with clinical benefit and in patients treated with osimertinib with or without LCT.

II. To determine modulation of genomic, proteomic and gene expression tumor profiles by induction osimertinib.

III. To explore osimertinib resistance mechanisms. IV. To determine the immunomodulatory effects of osimertinib plus LCT.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (LCT): Patients receive osimertinib orally (PO) once daily (QD) for 6-12 weeks. Patients then undergo surgery and/or radiation therapy daily for 5 consecutive days every week for up to 8 weeks. Patients continue osimertinib during and after radiation therapy. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

GROUP II (NO LCT): Patients receive osimertinib PO QD. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days, then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer
* Stage IIIB/IV or recurrent non-small cell lung cancer which is not amenable to curative intent therapy
* Patients must have one of the following:

  * NSCLC which harbors EGFR exon 19 deletion or L858R mutation. This subset of patients must be TKI naive; OR
  * NSCLC which harbors an EGFR T790M mutation that was acquired following progression on erlotinib, gefitinib or afatinib. This subset of patients must have not received prior third generation TKI
  * NOTE: EGFR mutation must be documented by a Clinical Laboratory Improvement Amendments (CLIA) certified test
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Candidate for local consolidation therapy to at least one site of disease
* Signed and dated written informed consent prior to admission to the study in accordance with International Council for Harmonization of Technical Requirements for Pharmaceuticals for Human Use (ICH)-Good Clinical Practice (GCP) guidelines and to the local legislation
* Ability to take pills by mouth
* Females of childbearing potential:

  * Must not be breast feeding
  * Must have a negative serum or urine pregnancy test
  * Must agree to use adequate contraception for a minimum of two weeks prior to receiving study medication until 3 months after discontinuation of the study medication

    * NOTE: Acceptable methods of contraception include total and true sexual abstinence, hormonal contraceptives that are not prone to drug-drug interactions (IUS levonorgestrel intra uterine system [Mirena], medroxyprogesterone injections [Depo-Provera]), copper-banded intra-uterine devices, and vasectomized partner. All hormonal methods of contraception should be used in combination with the use of a condom by their sexual male partner. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause)
* Women will be considered post-menopausal if they have been amenorrheic for the past 12 months without an alternative medical cause. The following age-specific requirements must also apply:

  * Women < 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of exogenous hormonal treatments. The levels of luteinizing hormone (LH) and follicle-stimulating hormone (FSH) must also be in the post-menopausal range (as per the institution)
  * Women >= 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of all exogenous hormonal treatments, or have had radiation-induced oophorectomy with the last menses > 1 year ago, or have had chemotherapy-induced menopause with > 1 year interval since last menses, or have had surgical sterilization by either bilateral oophorectomy or hysterectomy
* Non-sterilized males who are sexually active with a female partner of childbearing potential must use adequate contraception for the duration of the study and 3 month after the last dose of study medication. Adequate contraception methods include: birth control pills (e.g. combined oral contraceptive pill), barrier protection (e.g. condom plus spermicide, cervical/vault cap or intrauterine device), and abstinence. Patients should not father a child for 6 months after completion of the study medication. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing the study medication. If male patients wish to father children they should be advised to arrange for freezing of sperm samples prior to the start of the study medication
* Life expectancy >= 12 weeks
* To be eligible for randomization, patients must:

  * Meet all the inclusion criteria
  * Have no progression of disease after 6-12 weeks of osimertinib per RECIST 1.1. To assess for progressive disease patients must have the following imaging:

    * Either a positron emission tomography (PET)/computed tomography (CT) scan or a CT scan of the chest/abdomen/pelvis (or CT chest)
    * A CT scan or a magnetic resonance imaging (MRI) of the brain
  * Have target lesions (lesions that will be treated with LCT if the patient is randomized to that arm). Patients that have a complete response (CR) to front-line osimertinib (e.g. no visible disease to target) will continue to be followed for progression on study but will not be randomized

Exclusion Criteria:

* Previous treatment with osimertinib, or a 3rd generation EGFR TKI. NOTE: Patients who are receiving initial osimertinib (6-12 weeks) outside this study are not excluded
* Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4 (at least 3 week prior). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4
* Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 (with the exception of alopecia grade 2) at the time of starting study treatment
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib
* Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* Males and females of reproductive potential who are not using and effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry
* History of hypersensitivity of osimertinib (or active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib)
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirement
* Absolute neutrophil count < 1,500/mcL
* Platelet < 100,000/mcL
* Hemoglobin < 9.0 g/dL
* Total bilirubin > 1.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or > 3 times ULN in the presence of documented Gilbert's syndrome or liver metastases
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) > 2.5 times ULN or > 5 times ULN if liver metastases are present
* Creatinine clearance < 50 mL/min/1.73 m^2 by Cockcroft-Gault equation
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (corrected QT [QTc] using Fridericia's formula) > 470 msec
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiogram (ECG) e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 msec
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
* Patients will be excluded from randomization if they meet any of the following criteria:

  * Any of the exclusion criteria
  * Complete response to osimertinib or prior treatment to all visible lesions, such that no lesion is amenable to LCT. Note that patients can receive palliative radiation therapy prior to randomization to CNS lesions or those requiring urgent treatment (e.g. for pain or bleeding), but are only eligible for the study if they have one site amenable to further radiation therapy. In addition, these lesions will be counted towards the total number of metastases, and will also be counted as target lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From the start date of osimertinib assessed up to 4 years
  Will be estimated using Kaplan-Meier method. The stratified log-rank test will be performed to test the difference in time-to-event distributions between treatment groups. Stratified Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis and to estimate hazard ratios.

SECONDARY OUTCOMES:
Overall survival | From the treatment start date assessed up to 4 years
  Will be estimated using Kaplan-Meier method. The stratified log-rank test will be performed to test the difference in time-to-event distributions between treatment groups. Stratified Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis and to estimate hazard ratios.
Time to progression of target lesions | Up to 4 years
  Will be estimated using Kaplan-Meier method. The stratified log-rank test will be performed to test the difference in time-to-event distributions between treatment groups. Stratified Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis and to estimate hazard ratios.
Time to appearance of new metastases | Up to 4 years
  Will be estimated using Kaplan-Meier method. The stratified log-rank test will be performed to test the difference in time-to-event distributions between treatment groups. Stratified Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis and to estimate hazard ratios.
PFS in oligometastatic subgroup | Up to 4 years
  Will be estimated using Kaplan-Meier method. The stratified log-rank test will be performed to test the difference in time-to-event distributions between treatment groups. Stratified Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis and to estimate hazard ratios.
Incidence of adverse events | Up to 30 days post treatment
  Toxicity data related to the treatments will be summarized by frequency tables. The association between the types and severity of toxicity and the treatment groups will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Saumil Gandhi, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org